CLINICAL TRIAL: NCT07385599
Title: A First-in-Man (FIM) Study of the LAmbre™ II Left Atrial Appendage Occluder and Occluder Delivery System for Patients With Non-Valvular Atrial Fibrillation
Brief Title: FIM Study of the LAmbre™ II LAA Occluder in Non-Valvular AF Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LT-TS-154-2025-01
Record Dates: First submitted 2025-07-21; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF)
Keywords: Lifetech; FIM study; LAmbre™ II Left Atrial Appendage Occluder and Occluder Delivery System; LAmbre™ II; LAmbre™ II Left Atrial Appendage Occluder; Left Atrial Appendage Occluder; LAmbre™ II LAAO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LAmbre™ II Left Atrial Appendage Occluder and Occluder Delivery System (Experimental)
  Interventions: Device: LAmbre™ II Left Atrial Appendage Occluder and Occluder Delivery System

INTERVENTIONS:
Device: LAmbre™ II Left Atrial Appendage Occluder and Occluder Delivery System — To evaluate the preliminary safety and feasibility of the LAmbreTM II Left Atrial Appendage Occluder and the Occluder Delivery System in patients with non-valvular atrial fibrillation who are at increased risk for stroke and systemic embolism.

SUMMARY:
To evaluate the preliminary safety and feasibility of the LAmbreTM II Left Atrial Appendage Occluder and the Occluder Delivery System in patients with non-valvular atrial fibrillation who are at increased risk for stroke and systemic embolism.

DETAILED DESCRIPTION:
Worldwide, atrial fibrillation (AF) is the most common cardiac arrhythmia in adults. The prevalence of AF gradually increases with age; its prevalence is 0.5% ~ 0.8% among 45 ~ 59 year-olds, 1.8% ~ 5.9% among 60 ~ 69 year-olds, and 6.7% ~ 17.9% among > 79 year-olds. Thromboembolic complications are the leading cause of death and disability in patients with AF, with ischemic stroke being the most common complication. AF significantly increases the risk of stroke by 3- to 5-fold due to thrombosis caused by abnormal atrial beat. The overall risk of ischemic stroke in patients with AF is 20% ~ 30%, and strokes due to atrial fibrillation account for 20% of all strokes.

Oral anticoagulation (OAC) is the standard of care in the management of non-valvular atrial fibrillation for stroke prevention and is recommended in the USA and European guidelines. However, the use of warfarin, a traditional oral anticoagulant, requires frequent and careful monitoring to ensure adequate anticoagulation as well as to prevent over-anticoagulation. This necessitates frequent laboratory blood tests to maintain the International Normalization Ratio (INR), a measure of the efficacy of the warfarin regimen, which can lead to patient non-adherence. Sub-therapeutic INR does not prevent systemic embolization, and supratherapeutic INR is a risk for haemorrhage. Moreover, the impact of interactions with other drugs, diet, narrow therapeutic window, and other reasons limit the use of warfarin. Several studies have shown that in clinical practice anticoagulation is given to less than 50% ~ 60% of patients with indications and discontinuation rates of warfarin approach 33% per year. Non-vitamin K antagonist oral anticoagulants (NOAC) have been shown to have a non-inferiority or superior effect in stroke reduction compared to warfarin without the need for routine laboratory monitoring. However, due to the high cost of NOACs and the lack of stable and effective antagonists, treatment discontinuation rates of up to 20% have been reported, and there is still an absolute risk of bleeding of 2% to 3% per year. A safe and effective alternative to anticoagulation for the stroke prevention in AF is needed, as the bleeding risk of anticoagulation and the presence of patient refusal/non-adherence/intolerance to long-term anticoagulation.

For a majority of patients with atrial fibrillation, it appears that thrombus formation would be located in the Left atrial appendage (LAA). Previous studies have suggested that more than 90% of thrombi in patients with non-valvular atrial fibrillation (NVAF) are located in the LAA. Therefore, surgical and percutaneous techniques to occlude the LAA could be a solution to reduce the risk of ischemic stroke for patients with AF. Surgical ligation of the LAA during the mitral valve surgery can reduce the risk of stroke, however, it is difficult to completely close the LAA by surgical ligation. Studies evaluating the incidence of incomplete ligation of the LAA during mitral valve surgery have shown that TEE-detected incidence of incomplete LAA ligation is about 36%. The WATCHMAN device (Boston Scientific, Natick, Massachusetts) is the most studied percutaneous left atrial appendage closure (LAAC) device and has shown that safety and efficacy are non-inferior to warfarin. In the current 2023 ACC/AHA/ACCP/HRS Guideline, percutaneous LAAC has been classified as a Class 2a indication for stroke prevention in patients with AF, a moderate to high risk of stroke, and a contraindication to long-term oral anticoagulation due to a non-reversible cause. However, the implantation procedure does have adverse effects which include serious pericardial effusion, procedure-related ischemic stroke, and device embolization. Due to the anatomical diversity of the LAA, certain patients are not candidates for this device.

The LAmbre™ Left Atrial Appendage Closure System, manufactured by Lifetech Scientific (Shenzhen) Co. Ltd., is the first generation of LAmbre LAAO device which is CE-marked and is current approved in Hong Kong Hospital Authority for regular clinical use. It consists of a LAA Occluder and a Delivery System and is a percutaneous transcatheter device intended to prevent thrombus embolization from the left atrial appendage in patients who have nonvalvular atrial fibrillation. This self-expanding LAA Occluder consists of an umbrella and a cover connected by a central waist. Although the first generation of LAmbre LAAO device is associated with high implantation success rate of 99.7% and a relatively low major procedure-related complication rate of 2.9%, to better match the challenging anatomy of the LAA and to further improve procedural safety, the first generation of LAmbre LAA O device has been upgraded.

The LAmbre™ II Left Atrial Appendage Occluder is the second generation of LAmbre LAAO device which is used with the Occluder Delivery System to seal off the left atrial appendage to prevent thrombus embolization from the left atrial appendage (LAA) in patients who have non-valvular atrial fibrillation. As an upgraded version of the LAmbre™ Left Atrial Appendage Occluder, the LAmbre™ II Left Atrial Appendage Occluder has a number of modifications including: the connection of Umbrella and Cover has been changed from the welded connection to the snap connection, which allows the Umbrella and Cover to be freely combined; the PET Membrane of the Cover has been added with a PC coating; the shape of the Cover has been changed from conical shape to disc shape; the structure of the end of U-shaped hook has been changed from a single beam structure to a diamond shape structure; the material of the Cover changed from 72 NiTi wires to 144 NiTi wires This study is a first-in-man study aimed at preliminary assessing the safety and feasibility of the LAmbre™ II Left Atrial Appendage Occluder and Occluder Delivery System. The results of this study will be the basis for the design of subsequent confirmatory studies.

ELIGIBILITY:
Inclusion Criteria:

1. The patient age ≥18 years;
2. The patient has documented paroxysmal, persistent, or permanent non-valvular atrial fibrillation;
3. The patient has a CHA2DS2-VASc score of ≥ 2 in men and CHA2DS2-VASc score of ≥ 3 in women;
4. The patient is recommended for oral anticoagulation therapy, but there is an appropriate rationale for seeking a non-pharmacologic alternative to oral anticoagulation;
5. The patient is deemed suitable for LAA closure by the site investigator and a clinician not a part of the procedural team in the shared decision-making process, and this determination has been documented in the patient's medical record;
6. The patient is willing and able to comply with the required medication post-procedure and follow-up evaluations;
7. The patient (or his or her legally authorized representative) has been informed of the nature of the study, agrees to its provisions, and has been provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

Exclusion Criteria:

1. Pregnant or nursing patients and those who plan pregnancy during the study period. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days prior to the index procedure;
2. Patients with atrial fibrillation that is defined by a single occurrence, or that is transient or reversible (e.g., secondary to CABG, an interventional procedure, pneumonia, or hyperthyroidism);
3. Patients who require long-term anticoagulation for a condition other than atrial fibrillation;
4. Bleeding diathesis or coagulopathy;
5. Patients with rheumatic mitral valve disease, known severe mitral stenosis requiring surgical or percutaneous valve replacement, or existing mechanical valve prosthesis;
6. Active infection with bacteremia;
7. Known hypersensitivity or contraindication to aspirin, clopidogrel, heparin, any device material or component (nickel titanium, PET, polypropylene), and/or contrast sensitivity;
8. Prior atrial septal defect (ASD) or patient foramen ovale (PFO) surgical repair or implantation of closure device;
9. Left atrial appendage is obliterated and surgical ligated;
10. Underwent any cardiac or non-cardiac interventional or surgical procedure within 30 days prior to the procedure or planned to have the interventional or surgical procedure within 60 days after implant procedure (e.g., cardioversion, ablation, percutaneous coronary intervention, cataract surgery, etc.);
11. Recent (within 90 days prior to procedure) stroke, transient ischemic attack, or myocardial infarction;
12. New York Heart Association Class IV;
13. Patients with severe renal failure (estimated glomerular filtration rate<30 ml/min/1.73m2);
14. Known asymptomatic carotid artery disease with>70% diameter stenosis OR symptomatic carotid disease (>50% diameter stenosis with ipsilateral stroke or TIA). Subjects with prior carotid endarterectomy or carotid stent placement may be enrolled, provided that known diameter stenosis is <50%;
15. Life expectancy is less than 1 year;
16. Current participation in another investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
The primary effective endpoint is closure success | 12 months post-procedure.
  Defined as complete LAA closure or peri-device residual leak ≤ 3 mm measured by TEE.
The primary safety endpoint is major peri-procedural complications | Within 7 days following the implant procedure or by hospital discharge
  Including cardiac perforation, pericardial effusion with tamponade or requiring drainage, device embolization, death, ischemic stroke, systemic embolism, and major vascular complications occurring within 7 days following the implant procedure or by hospital discharge, whichever is later.

SECONDARY OUTCOMES:
Major adverse events | Evaluated within 7 days following the implant procedure or by hospital discharge and 30 days and 3, 6, 12 months post-procedure
  Defined as death, stroke, systemic embolism, pericardial effusion with tamponade or requiring drainage, device embolization, and major bleeding (BARC defined 3 or 5)
Closure success | Evaluated at 30 days and 3, 6 months post-procedure
  Assessed by TEE or cardiac computed tomography
Rate of bleeding complications | Evaluated within 7 days following the implant procedure or by hospital discharge, 30 days and 3, 6, 12 months post-procedure
  Evaluated as major bleeding (BARC Type 3 or 5) and minor bleeding (BARC type 2)
Cardiovascular death | Evaluated within 7 days following the implant procedure or by hospital discharge, 30 days and 3, 6, 12 months post-procedure
  (cardiovascular and/or unexplained cause)
Rate of ischemic stroke and systemic embolization | Evaluated within 7 days following the implant procedure or by hospital discharge, 30 days and 3, 6, 12 months post-procedure
Technical success rate | Evaluated immediately after the procedure
  Defined as successful delivery and release of study device with acceptable device position and stability, and closure success
Procedural success rate | Evaluated at 7 days following the implant procedure or by hospital discharge, whichever comes later
  Defined as technical success without major peri-procedural complications
Device-related thrombosis | Evaluated at 30 days and 3, 6, 12 months post-procedure
  Defined as the detection of thrombus adherent to the left atrial side of the device by TEE or cardiac computed tomography
Occluder Delivery System related complication | Evaluated immediately after the procedure and within 7 days following the implant procedure or by hospital discharge
Performance Assessment of the Occluder Delivery System | Evaluated during the procedure
  Including accuracy, flexibility, pushability, withdrawal of delivery system (Grade I-V, V represents the best).
Performance Assessment of the Occluder Delivery System: Puncture success | Evaluated during the procedure
  Defined as the successful puncture of the oval fossa region of the interatrial septum under fluoroscopy or TEE guidance, without changing the puncture needle or puncture site. The delivery sheath and dilator are then successfully advanced into the left atrium.

CONTACTS AND LOCATIONS:
Overall Officials: Kent CY So, Professor, Principal Investigator — Prince of Wales Hospital, Chinese University of Hong Kong, HKSAR
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, HKSAR, Shatin, Hong Kong